CLINICAL TRIAL: NCT00725543
Title: Remicade Therapy in Ankylosing Spondylitis: Investigation of Real Life Regimen in Austria Over 9 Consecutive Infusions
Brief Title: Investigation of 9 Consecutive Remicade Infusions in Ankylosing Spondylitis in Austria (Study P04044)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P04044
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Remicade: Subjects with AS with severe axial symptoms and elevated serological markers of inflammatory activity will receive Remicade induction therapy consisting of 3 Remicade infusions in weeks 0, 2, and 6 given in specialized centers. Maintenance therapy will consist of another maximal 6 infusions given in doses and intervals due to discretion of physicians. Whole observation period cannot exceed 102 weeks per subject if the maximal therapy interval of 16 weeks as defined in Summary of Product Characteristics (SPC) is taken into consideration.
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Remicade induction therapy consists of 3 infusions given at weeks 0, 2, and 6 in specialized centers. Maintenance therapy will consist of a maximum of 6 infusions given in doses and intervals due to discretion of physicians.
  Other Names: Remicade; SCH 215596

SUMMARY:
This is a prospective, open-label, 1-arm, multicenter observational study to determine the dose and time span of Remicade between infusions for ankylosing spondylitis (AS).

DETAILED DESCRIPTION:
This study population was chosen from a non-probability sample.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ankylosing spondylitis with severe axial symptoms and elevated serological markers of inflammatory activity.

Exclusion Criteria:

* Subjects with tuberculosis or other severe infections such as sepsis, abscesses, and opportunistic infections.
* Subjects with moderate or severe heart failure (New York Heart Association (NYHA) class III/IV).
* Subjects with a history of hypersensitivity to Remicade or to other murine proteins, or to any of the excipients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with AS will receive Remicade induction therapy at specialized centers.
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2004-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Remicade: Remicade induction therapy consisted of 3 infusions (5 mg/kg) in weeks 0, 2, and 6 given in specialized centers. Maintenance therapy consisted of a maximum of 6 infusions (5 mg/kg) given in doses and intervals at the discretion of physician. The observation period could not exceed 102 weeks per participant if the maximal therapy interval of 16 weeks as defined in Summary of Product Characteristics (SPC) was taken into consideration.
Period: Overall Study
Arm/Group | Remicade
Started | 358
Completed | 205 (Completed was defined as the number of participants who received 9 consecutive Remicade infusions.)
Not Completed | 153
Not completed — Adverse Event | 10
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 10
Not completed — Physician Decision | 5
Not completed — Lost to Follow-up | 4
Not completed — Non-compliance | 2
Not completed — Other | 119

BASELINE CHARACTERISTICS:
Arm/Group | Remicade
Number analyzed (Participants) | 358
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.08 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 260

OUTCOME MEASURES:

1. Primary Outcome: Mean Time Interval Between Remicade Infusions in Participants During Maintenance Treatment Following Induction Therapy
Time Frame: Maximum of 24 months
Population: Remicade-naive participants who received Remicade induction therapy and subsequent maintenance therapy during the observational study.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Remicade
Number analyzed (Participants) | 165
Days
  Infusion 3/4 (n=165) | 56.10 (10.97)
  Infusion 4/5 (n=165) | 60.62 (25.58)
  Infusion 5/6 (n=159) | 57.91 (8.11)
  Infusion 6/7 (n=154) | 59.39 (15.91)
  Infusion 7/8 (n=152) | 59.52 (17.67)
  Infusion 8/9 (n=143) | 60.36 (17.96)

2. Primary Outcome: Median Time Interval Between Remicade Infusions in Participants During Maintenance Treatment Following Induction Therapy
Time Frame: Maximum of 24 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Remicade
Number analyzed (Participants) | 165
Days
  Infusion 3/4 (n=165) | 57.00 [26.00 to 141.00]
  Infusion 4/5 (n=165) | 57.00 [19.00 to 340.00]
  Infusion 5/6 (n=159) | 57.00 [15.00 to 84.00]
  Infusion 6/7 (n=154) | 57.00 [29.00 to 176.00]
  Infusion 7/8 (n=152) | 57.00 [42.00 to 211.00]
  Infusion 8/9 (n=143) | 57.00 [30.00 to 157.00]

3. Primary Outcome: Mean Dose of Remicade in Participants Receiving Induction Therapy and Subsequent Maintenance Therapy
Time Frame: Maximum of 24 months.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams/kilograms (mg/kg)
Arm/Group | Remicade
Number analyzed (Participants) | 165
milligrams/kilograms (mg/kg)
  Infusion 1 (n=163) | 4.37 (0.93)
  Infusion 2 (n=164) | 4.39 (0.90)
  Infusion 3 (n=164) | 4.43 (0.88)
  Infusion 4 (n=165) | 4.42 (0.89)
  Infusion 5 (n=165) | 4.44 (0.87)
  Infusion 6 (n=160) | 4.47 (0.87)
  Infusion 7 (n=154) | 4.54 (0.91)
  Infusion 8 (n=152) | 4.59 (0.94)
  Infusion 9 (n=143) | 4.67 (0.93)

4. Primary Outcome: Median Dose of Remicade in Participants Receiving Induction Therapy and Subsequent Maintenance Therapy
Time Frame: Maximum of 24 months.
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Remicade
Number analyzed (Participants) | 165
mg/kg
  Infusion 1 (n=163) | 4.60 [2.35 to 7.02]
  Infusion 2 (n=164) | 4.62 [2.35 to 7.02]
  Infusion 3 (n=164) | 4.62 [2.38 to 7.02]
  Infusion 4 (n=165) | 4.62 [2.32 to 7.02]
  Infusion 5 (n=165) | 4.62 [2.44 to 7.02]
  Infusion 6 (n=160) | 4.66 [2.44 to 7.02]
  Infusion 7 (n=154) | 4.68 [2.41 to 7.69]
  Infusion 8 (n=152) | 4.71 [2.35 to 7.69]
  Infusion 9 (n=143) | 4.71 [2.33 to 7.69]

5. Primary Outcome: Mean Remicade Dose Per Participant
Time Frame: Maximum of 24 months
Population: Remicade-naive participants who were exposed to Remicade during the observational study.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Remicade
Number analyzed (Participants) | 348
mg/kg | 4.53 (0.84)

6. Primary Outcome: Median Remicade Dose Per Participant
Time Frame: Maximum of 24 months
Population: Remicade-naive participants who were exposed to Remicade during the observational study.
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Remicade
Number analyzed (Participants) | 348
mg/kg | 4.75 [1.98 to 7.02]

ADVERSE EVENTS:
Arm/Group | Remicade
Serious Adverse Events (participants affected / at risk) | 4/358
Other Adverse Events (participants affected / at risk) | 0/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remicade (N=358)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Infusion Related Reaction (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Lymph Node Tuberculosis (Infections and infestations) | 1 (1)
Mixed Oligo-astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No